CLINICAL TRIAL: NCT00107367
Title: A Phase I/II Study Utilizing the Zeiss INTRABEAM System for the Treatment of a Resected Solitary Brain Metastasis
Brief Title: Radiation Therapy in Treating Patients Who Are Undergoing Surgery to Remove a Metastatic Brain Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Robert Weil, Cleveland Clinic Taussig Cancer Center
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000378144; CCF-IRB-7003; CCF-510K; CCF-K992577; CCF-CTSRC-1065
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-07

CONDITIONS: Metastatic Cancer
Keywords: tumors metastatic to brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms

INTERVENTIONS:
Procedure: conventional surgery
Radiation: intraoperative radiation therapy

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers radiation directly to the area where a tumor was surgically removed may kill any remaining tumor cells and cause less damage to normal tissue.

PURPOSE: This phase I/II trial is studying radiation therapy to see how well it works in treating patients who are undergoing surgery to remove a metastatic brain tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 1-year local control rate in patients undergoing resection of a solitary brain metastasis comprising intraoperative radiotherapy using the INTRABEAM® system.

Secondary

* Determine the survival of patients treated with this therapy.
* Determine distant recurrence of disease in patients treated with this therapy.
* Determine the toxicity of this therapy in these patients.
* Determine the quality of life of patients treated with this therapy.

OUTLINE: This is a nonrandomized study.

Patients undergo surgical resection of a brain metastasis. Patients then undergo intraoperative radiotherapy using the INTRABEAM® system.

Quality of life is assessed at baseline and then every 3 months for 2 years.

Patients are followed within 48 hours after surgery, at 1 and 3 months, and then every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 31-62 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed supratentorial solitary brain metastasis by enhanced MRI or CT scan

  * Resectable disease
  * Histological evidence of metastatic carcinoma by intraoperative pathology
* No primary lymphoma, germ cell carcinoma, or small cell lung cancer

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 3 months

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No uncontrolled hypertension
* No unstable angina pectoris
* No uncontrolled dysrhythmias

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious infection
* No other medical illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior temozolomide or polifeprosan 20 with carmustine implant (Gliadel® wafer) for brain metastasis

Endocrine therapy

* Not specified

Radiotherapy

* No prior brain radiotherapy of any kind, including local or whole brain external beam radiotherapy, brachytherapy, or stereotactic radiosurgery
* No concurrent external beam radiotherapy to the brain
* Not planning adjuvant whole brain radiotherapy after study therapy

Surgery

* Not specified

Other

* No other prior conventional or investigational local or systemic agents for brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2004-04; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Local control rate as measured by MRI with contrast at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Weil, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Weil RJ, Mavinkurve GG, Chao ST, Vogelbaum MA, Suh JH, Kolar M, Toms SA. Intraoperative radiotherapy to treat newly diagnosed solitary brain metastasis: initial experience and long-term outcomes. J Neurosurg. 2015 Apr;122(4):825-32. doi: 10.3171/2014.11.JNS1449. Epub 2015 Jan 23. PMID 25614945